CLINICAL TRIAL: NCT01248182
Title: Bone to Skin Thickness Study: Obese Versus Normal Population
Status: Terminated | Type: Observational
Why Stopped: Study was terminated by investigator
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009-0059
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Fracture
Keywords: acetabular fracture; pelvic ring injury
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the bone to skin depth for groups of lean, obese and morbidly obese patients. This information will be potentially helpful with implant design for obese and lean patients.

DETAILED DESCRIPTION:
This study will examine pelvic CT scans of injured patients to determine skin thickness in several distinct regions important in orthopedic surgery. All patients admitted to the University of Mississippi Medical Center with a pelvic ring injury or acetabular fracture obtain a pelvic CT scan as a standard part of patient evaluation. The CT scans attempt to encompass the entire soft tissue sleeve from the skin edge to the pelvic bones. Several landmarks described below have been described to measure important surgical sites where obesity is problematical. Therefore this study is an attempt to quantify the size of the soft tissue envelope in patients

However, patients who are markedly obese may be too large for the entire soft tissue sleeve to be imaged with the CT scan. The second part of the study then is to validate the CT scan measurements obtained using clinical measurements. The clinical measurements will be obtained during operative management of displaced pelvic ring injuries and/or acetabular fractures. During surgical exposure, a measuring tape will be used to measure the soft tissue thickness in those areas corresponding to the CT scan measurements. These measures will be compared to validate the effectiveness of CT scan measurements to accurately document the soft tissue dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Anyone admitted to the University of Mississippi Medical Center with a pelvic ring or acetabular injury

Exclusion Criteria:

* Those not fitting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pelvic ring injury or acetabular fracture
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Graves, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States